CLINICAL TRIAL: NCT03380832
Title: Vestibular Perception and Action
Brief Title: Motion Perception in Individuals With Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Faisal_Karmali@MEEI.HARVARD.EDU, Principal Investigator, Massachusetts Eye and Ear Infirmary
Other Study IDs: 196245
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes for at least 10 years: This is an observational study in which we will quantify vestibular thresholds in individuals who have had type 2 diabetes for at least 10 years. Normative data has recently been published and subjects with diabetes will be compared to a model that includes age effects.

SUMMARY:
Is the ability to perceive motion altered by diabetes? The investigators are measuring motion perception using a technique called vestibular thresholds. Subjects will undergo 3 hours of testing in which they sit in a chair that makes small movements and report their perception of motion. The investigators are currently looking for individuals who have had type 2 diabetes for at least 10 years.

DETAILED DESCRIPTION:
Previous studies have found that individuals with diabetes fall more frequently, have less stable posture, and have reduced motion and touch sensation in the lower extremities. This study will examine whether vestibular sensation is also affected by diabetes.

This study is observational because measurements will be made without the application of an intervention. The same measurement protocol was applied to a large group of normal subjects, and this published data will serve as normative controls.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 10 years
* Under 250 pounds

Exclusion Criteria:

* Medications not to be used include: Ambien (Zolpidem), Antivert, Bonine (Meclizine), Ativan (Lorazepam), Benadryl (diphenhydramine), Dalmane (Flurazepam), Dramamine, Doral (Quazepam), Fiorinal, Fiorcet (Butalbital), Halcion (Triazolam), Klonopin (Clonazepam), Librium, Librax (Chlordiazepoxide), Nembutal (Pentobarbital), Phenergan (Promethazine), Placidyl (Ethchlorvynol), Prosom (Estazolam), Restoril (Temazepam), Seconal (Secobarbital), Serax (Oxazepam), Transderm Scopes Patch, Vontrol (Diphenidol), Xanax (Alprazolam).
* Individuals meeting the following criteria will be excluded: a) a history of head trauma, b) posterior fossa pathology, c) a well-defined otologic diagnosis (e.g., Benign Paroxysmal Positional Vertigo (BPPV), Meniere's disease, superior canal dehiscence, etc., unilateral or bilateral vestibular hypofunction) d) a recent history of seizures e) any other major neurologic (e.g., Parkinson's, Multiple Sclerosis, dementia, epilepsy, cerebellar ataxia, stroke, recent concussion, etc.) disorder, f) any major psychiatric (e.g., panic disorder, psychosis, etc.) disorder, and g) any other severe health problem (heart disease, pulmonary disease, cancer, etc.).
* Due to nauseogenic nature of some motions and to protect fetus and mother, pregnant women will also be excluded from this study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Vestibular threshold | 3 hours
  Vestibular thresholds are measured while subjects sit in a chair that makes small motions in a variety of directions. After each motion, subjects press a button to report their perceived direction (e.g., did I rotate to the left or the right). The size of the motions is adjusted based on subject responses to find the level at which they get approximately 80% of responses correct.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Karmali, PhD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided